CLINICAL TRIAL: NCT06764225
Title: Effects of Low-Sodium Substitute Salt on Death, Heart Failure Hospitalization, Heart Failure Emergency Department Visits, and Quality of Life in Patients With Heart Failure: A Multicenter, Double-Blind, Randomized Controlled Trial
Brief Title: Effects of Low-Sodium Salt on Death, HF Hospitalization/ Emergency Department Visits and Quality of Life in HF Patients
Acronym: RESCUE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Health Research Center (Other)
Collaborators: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RESCUE-HF
Record Dates: First submitted 2024-12-24; First posted 2025-01-08 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Dietary Sodium Intake
Keywords: low-sodium substitute salt
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-sodium substitute salt (Experimental): Low-sodium substitute salt
  Interventions: Other: low-sodium substitute salt
- Regular Salt (No Intervention): Regular Salt

INTERVENTIONS:
Other: low-sodium substitute salt — This study specifically customized sodium reducing substitute salts with a sodium chloride content not exceeding 62% and without the addition of potassium chloride.
  Arms: Low-sodium substitute salt

SUMMARY:
This study aims to investigate whether using a low-sodium substitute salt can help improve outcomes for patients with heart failure. Specifically, it will examine if the low-sodium substitute salt can reduce death rates, hospital readmissions, and emergency visits, as well as improve the quality of life for these patients.

DETAILED DESCRIPTION:
The study will involve multiple centers and use a randomized, double-blind, controlled design, where participants will be randomly assigned to either the intervention group (who will use the low-sodium substitute salt ) or the control group (who will use regular salt). Participants will be followed up for at least a year, assessing outcomes including all cause mortality, heart failure hospitalizations, emergency visits, and changes in quality of life as measured by a questionnaire.

Eligible participants will be between 18 and 75 years old, have been hospitalized for heart failure in the past year, and have stable heart failure. The study will exclude individuals with severe heart failure, uncontrolled health conditions, or other factors that may interfere with participation.

The main goals are to determine if reducing sodium intake through the low-sodium substitute salt leads to better health outcomes in heart failure patients over a year. Participants will be followed up at 3, 6, 9, and 12 months.

This research will help provide evidence for whether a simple dietary change, like using a low-sodium substitute salt , can make a meaningful difference in managing heart failure

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years;
2. Hospitalized due to heart failure in the past year;
3. NYHA functional class II-III;
4. Echocardiographic evidence of LVEF < 40% within the past 6 months;
5. Receiving guideline-directed medical therapy for heart failure;
6. Stable heart failure status, defined as heart failure stability for more than 4 weeks, with no increase in diuretic dose within the past 4 weeks;
7. Having a primary caregiver and frequently dining together at home;
8. Consuming commercially processed food no more than once a week;
9. Providing written informed consent.

Exclusion Criteria:

1. End-stage heart failure;
2. Hospitalization due to cardiovascular causes within the past month;
3. Uncorrected hyponatremia (Na < 130 mmol/L);
4. Dialysis-dependent patients, or eGFR < 20 mL/min/1.73m²;
5. Uncontrolled hyperglycemia, with fasting blood glucose > 16 mmol/L;
6. Malignant cancer patients with a life expectancy of less than 1 year;
7. Conditions that, in the investigator's opinion, may interfere with adherence to the protocol, such as habitual reliance on takeout meals or dining at company cafeterias;
8. Planned hospitalization during the study period;
9. Unexplained weight loss greater than 5 kg in the past year;
10. The subject or family members have concerns about using the salt substitute in this study, or are planning for pregnancy, pregnant, or breastfeeding;
11. Another family member is already participating in this study;
12. The subject or family members are participating in other interventional clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1301 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of pairwise comparisons with wins of a composite endpoint including 1-year death, the number of HF hospitalizations/emergency visits, time to the first HF hospitalization/emergency visit, and the change in quality of life at 12 months | From enrollment to the end of follow-up at 1 year
  Clinical benefit, a composite of all cause death, the number of HFHs/emergency visits, time to the first HFH/emergency visit, and the change in quality of life (Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) )at 1 year. All patients randomized to low-sodium group are compared to those randomized to control group within strata. For any two patients, a patient will win, i.e. achieve a better clinical outcome, as determined by assessing the following criteria sequentially, stopping when an advantage for either patient is shown:
  1. Death: death is worse than no death; earlier death is worse; tied if not possible to determine.
  2. Number of HF hospitalizations/emergency visits,: more HFHs/emergency visits is worse; tied, if same number.
  3. Time to first HFH/emergency visit: earlier HFH/emergency visit is worse; tied, if not possible to determine.
  4. KCCQ-12 at 1 year: Higher KCCQ-12 is better. The KCCQ-12 ranges from 0 to 100, where a higher score reflects a better outcome.

SECONDARY OUTCOMES:
1-year all-cause mortality | From enrollment to the end of follow-up at 1 year
The number of heart failure hospitalizations/emergency visits within 1 year | From enrollment to the end of follow-up at 1 year
Time from randomization to the first heart failure hospitalization/emergency visit | From enrollment to the end of follow-up at 1 year
Cardiovascular mortality within 1 year | From enrollment to the end of follow-up at 1 year
Change in heart failure quality of life score (KCCQ) | From enrollment to the end of follow-up at 1 year
  The KCCQ-12 ranges from 0 to 100, where a higher score reflects a better outcome.
Change in frailty score for heart failure (FRIED scale) | From enrollment to the end of follow-up at 1 year
  The FRIED scale assesses frailty in older adults based on five criteria: weight loss, exhaustion, weakness, slowness, and low activity. Frailty is classified as non-frail (0), pre-frail (1-2), or frail (≥3), predicting risks like falls, hospitalization, and mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided